CLINICAL TRIAL: NCT00246922
Title: A Long-term Study of APTA-2217 in Adult Patients With Bronchial Asthma
Brief Title: Long-term Study of Safety and Efficacy of Roflumilast in Japanese Patients With Bronchial Asthma (20 to 71 y) (APTA-2217-07)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: APTA-2217-07
Record Dates: First submitted 2005-10-31; First posted 2005-11-01 (Estimated); Last update posted 2016-12-02 (Estimated); Status verified 2016-09

CONDITIONS: Bronchial Asthma
Keywords: Asthma; Roflumilast; phosphodiesterase 4 inhibitor
MeSH Terms: conditions — Asthma | interventions — Roflumilast

INTERVENTIONS:
Drug: Roflumilast

SUMMARY:
The aim of this long-term study is to investigate the effect of roflumilast (APTA-2217) on the long-term safety in patients with asthma, who completed the 24-week evaluation of study APTA-2217-05. Roflumilast will be administered orally once daily. The present study consists of a 28 weeks treatment period, and is the extension of the 24-week study APTA-2217-05 (registered study). The study will provide further long-term safety and efficacy data of roflumilast.

ELIGIBILITY:
Main inclusion criteria:

* Patients with asthma disease
* Written informed consent
* Patients who completed the 24-week evaluation of study APTA-2217-05

Main exclusion criteria:

* % FEV1.0 < 60% at both 18 weeks and 24 weeks measurements during APTA-2217-05
* Patients with poorly controlled asthma between informed consent day and study starting day: need for oral or intravenous steroid therapy, hospitalization or any emergency visit, PEF value worsened for 2 or more consecutive days
* Serious diseases

Ages: 20 Years to 71 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2004-12; Primary Completion 2007-01 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Long-term safety after 28 weeks treatment of Roflumilast at (total 52 weeks, 24 weeks of study APTA-2217-05 followed by 28 weeks) .

SECONDARY OUTCOMES:
Efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AstraZeneca, Study Director — AstraZeneca
Locations (1):
- Nycomed Japan and Mitsubishi Tanabe Pharma Corporation, Osaka, Japan

REFERENCES:
- See also: APTA-2217-07-RDS-2009-01-16.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4467&filename=APTA-2217-07-RDS-2009-01-16.pdf